CLINICAL TRIAL: NCT04710953
Title: Comparison of Effectiveness Between Continuous Positive Airway Pressure (CPAP) and Hyperbaric Chamber Ventilation for the Patients of High Altitude Pulmonary Edema (HAPE) When Given in Addition to Standard of care-a Randomized Control Trial
Brief Title: Comparison of CPAP and Gamow Bag Ventilation to Treat HAPE
Acronym: CPAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: sultan mehmood kamran (Other)
Collaborators: Pak Emirates Military Hospital (Other); HALMARC (Unknown)
Responsible Party: Sponsor-Investigator, sultan mehmood kamran, Classified Medical specialist, UNICEF
Organization: UNICEF (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HALMARC
Record Dates: First submitted 2021-01-10; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: High Altitude Pulmonary Edema
Keywords: high altitude; CPAP; hyperbaric chamber; Gamow bag; AMS
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Intervention Model Description: Study Design: Randomised control trial Settings: Posts more than 8000 feet (2400m) where Medical officer is available Study Duration: 01 year after the study is approved Sampling Technique: Non probability consecutive sampling Distribution of patients in to two groups (Gp A and Gp B) by consecutive sampling Group "A" will be given CPAP in addition to standard of care and Group B will be offered Gamow bag in addition to standard of care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CPAP arm (Experimental): In addition to standard of care, CPAP will be provided at high altitude posts where Gamow bag is not available and all patients of HAPE will be given CPAP when evacuation/descent is either not possible or delayed due to weather conditions.
  Interventions: Device: Continuous positive airway pressure machine
- Gamow bag arm/hyperbaric chamber (No Intervention): Posts where Gamow bag would be available, the patients of HAPE will be given standard of care and will be asked to lie inside Gamow bag inflated at 2 Psi for several hours to simulate a descent of 1500 meters when evacuation/descent is either not possible or delayed due to weather conditions.

INTERVENTIONS:
Device: Continuous positive airway pressure machine — CPAP device set at 6-8cmH2O for several hours
  Other Names: CPAP-REMstar pro (system one 60 series)
  Arms: CPAP arm

SUMMARY:
High altitude pulmonary edema (HAPE) is mostly treated with supplemental oxygen, nifedipine 30mg twice a day, rest, limiting cold exposure and descent (simulated or actual) Gamow Bag provides simulated descent and buy time for actual descent. CPAP is claimed to be effective in many case reports to treat HAPE temporarily until actual descent is taken place. This study aims to evaluate the role of CPAP in treating HAPE at those high altitude stations where Gamow bag is not available and immediate descent is not possible.

DETAILED DESCRIPTION:
Background:

Swenson described HAPE in 2002, as a form of hydrostatic acute pulmonary edema with an alteration of alveolar-capillary permeability. Overall prevalence of AMS is 10-20% while incidence of HAPE, HACE or mixed incidence is 2-3%. Highest reported incidence of HAPE among Indian soldiers climbing to Siachen glacier is 15.5%. At 1500-2400m, A series of 52 patients admitted for HAPE over a period of 9 years was reported in literature..

Scientific rationale:

Positive pressure has been used to increase altitude tolerance since the 1940s under simulated altitudes. PEEP applied via face mask increased SpO2 and decreased AMS symptoms. CPAP was used after ascent to 3205 m on Mount Cook in New Zealand where it improved SpO2 and reduced symptoms of HAPE. A CPAP helmet providing 15 cmH20 CPAP improved SpO2 in a single HAPE patient (at 5300 m) from 56% to 74%.-1st case report. A study at Thorang La pass (5416 m) in October 2010 in the Nepal Himalaya found that nasal continuous positive airway pressure (CPAP) is useful as an additional modality to treat presumed high altitude pulmonary edema (HAPE)- 2nd case report.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Age 18-45 years
* Previously fit and no comorbids
* Suspected HAPE

  --arrived in the past 01 week on the post
* Expected evacuation from post more than 8 hours

Exclusion Criteria:

* Symptoms suggest acute infective etiology.
* Symptoms after one week of stay at HA
* Altered mental status.
* Disturbed balance
* Visual impairment
* Severe headache
* A speedy evacuation to a lower height is available

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Resolution of HAPE | 8 hours
  No dyspnea at rest, 2. RR < 20 3. Pulse < 100 4. O2 sat > 90% 5. Chest clears to auscultation
  Pulse < 100 O2 sat > 90% CheComplete resolution of HAPE symptoms RR < 20 Pulse < 100 O2 sat > 90% Chest clear to auscultation complete resolution of HAPE symptoms with RR < 20, Pulse < 100, O2 saturation > 92% and chest clear to auscultation

SECONDARY OUTCOMES:
Partial improvement in HAPE features | 8 hours
  Partial improvement in symptoms and signs as measured by at least one grade improvement in MMRC score, at least 25 percent improvement in all or some of the vital signs or oxygen saturations

CONTACTS AND LOCATIONS:
Overall Officials: Imran Fazal, FCPS, Study Director — Pak Emirates Military Hospital Rawalpindi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gabry AL, Ledoux X, Mozziconacci M, Martin C. High-altitude pulmonary edema at moderate altitude (< 2,400 m; 7,870 feet): a series of 52 patients. Chest. 2003 Jan;123(1):49-53. doi: 10.1378/chest.123.1.49. PMID 12527602
- [Result] Johnson PL, Johnson CC, Poudyal P, Regmi N, Walmsley MA, Basnyat B. Continuous positive airway pressure treatment for acute mountain sickness at 4240 m in the Nepal Himalaya. High Alt Med Biol. 2013 Sep;14(3):230-3. doi: 10.1089/ham.2013.1015. PMID 24067184
- [Result] Koch RO, Hinterhuber L, Faulhaber M, Gatterer H, Graupner S, Muenzel K, Burtscher M. A successful therapy of high-altitude pulmonary edema with a CPAP helmet on Lenin Peak. Clin J Sport Med. 2009 Jan;19(1):72-3. doi: 10.1097/JSM.0b013e3181915cce. No abstract available. PMID 19124989
- [Result] Ginosar Y, Malhotra A, Schwartz E. High altitude, continuous positive airway pressure, and obstructive sleep apnea: subjective observations and objective data. High Alt Med Biol. 2013 Jun;14(2):186-9. doi: 10.1089/ham.2012.1085. PMID 23795742